CLINICAL TRIAL: NCT02494466
Title: The Effects on Airway Reactivity of the Use of Preoperative Montelukast Sodium
Brief Title: Preoperative Use of Montelukast Sodium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: GK6
Record Dates: First submitted 2015-05-05; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Airway Reactivity
Keywords: Airway Resistance; montelukast sodium; laryngeal mask airway
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group E (n=10) (Active Comparator): Patients with high Ig E levels
  Interventions: Drug: montelukast sodium
- Group C (n=10) (Active Comparator): Patients with normal Ig E levels
  Interventions: Drug: montelukast sodium
- Group M (n=10) (Active Comparator): Patients who would be administered with 4mg PO MS 10 days before surgery because of high IgE
  Interventions: Drug: montelukast sodium

INTERVENTIONS:
Drug: montelukast sodium — 4 mg peroral Montelukast Sodium, 10 days before surgery because of high IgE.

SUMMARY:
Supraglottic airway equipment used during anaesthesia application can lead to airway reactivity or even larynx spasm in sensitive children.

Montelukast Sodium, used in asthma treatment, is a cysteinyl leukotriene Type 1 antagonist which reduces leukotriene C4, leukotriene D4 and leukotriene E4 synthesis. The use of Montelukast Sodium in airway reactivity is known to reduce the need for bronchodilator and corticosteroids.

DETAILED DESCRIPTION:
The study will comprise 30 american society of anesthesiology (ASA) I-III patients, aged 4-8 years, undergoing inguinal hernia surgery. Patients will exclude if receiving asthma treatment, if they had upper respiratory tract infection in the last week and if the laryngeal mask airway (LMA) could not be placed at a single attempt.

Patients will be separated into 3 groups as Group E (n=10) with high immunoglobulin E (IgE), Group C (n=10) with normal IgE and Group M (n=10) who were administered with 4mg peroral Montelukast Sodium, 10 days before surgery because of high IgE.

With spontaneous breathing after anaesthesia induction, a classic LMA will be placed. Anaesthesia will be maintained with a mixture of 1.3 minimum alveolar concentration (MAC) sevoflurane 500%2 - N2O. At 5-minute intervals, oxygen saturation (sPO2), End-Tidal carbon dioxide, Heart Rate, tidal volume (VT), respiratory rate (f) and peak airway pressure (PAP) will be monitored and coughing, apnea, laryngospasm , bronchospasm, desaturation and need for steroids will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing inguinal hernia surgery

Exclusion Criteria:

* If receiving asthma treatment,
* If they had URTI in the last week and
* If LMA could not be placed at a single attempt.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with bronchospasm as a Measure of airway reactivity | during the operation
Number of Participants with laryngospasm as a Measure of airway reactivity | during the operation
Number of Participants with apnea | during the operation

SECONDARY OUTCOMES:
amount of applied steroids | during the operation
  steroids can prevent airway reactivity symptoms
peak airway pressures as a measurement of airway reactivity | during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Bakan, MD, Study Chair — Unraniye training and research hospital
Locations (1):
- Gulsah Karaoren, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Casares-Alonso I, Cano-Garcinuno A, Blanco-Quiros A, Perez-Garcia I. Anti-asthmatic prescription variability in children according to age. Allergol Immunopathol (Madr). 2015 Jul-Aug;43(4):383-91. doi: 10.1016/j.aller.2014.05.010. Epub 2014 Oct 23. PMID 25444114
- [Result] Bush A. Montelukast in paediatric asthma: where we are now and what still needs to be done? Paediatr Respir Rev. 2015 Mar;16(2):97-100. doi: 10.1016/j.prrv.2014.10.007. Epub 2014 Dec 12. PMID 25499571